CLINICAL TRIAL: NCT02820246
Title: NutritionDay in Worldwide Hospitals: A Cross-sectional Registry
Brief Title: NutritionDay in Worldwide Hospitals: An International Audit and Registry on Nutrition and Outcome
Acronym: nutritionday
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: European Society for Clinical Nutrition and Metabolism (Other); Austrian Society for Clinical Nutrition (Other)
Responsible Party: Principal Investigator, Michael J. Hiesmayr, Professor of Anesthesia and Intensive Care, Medical University of Vienna
Other Study IDs: 407/2005
Record Dates: First submitted 2016-06-27; First posted 2016-06-30 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Malnutrition
Keywords: nutrition assessment; nutrition therapy; nutrition surveys; patient outcome assessment; outcome and process assessment; benchmarking; risk assessment; scoring system
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Status; Food Service, Hospital; Enteral Nutrition; Parenteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- hospitalised patients: all patients present in a hospital ward during the morning shift
  Interventions: Other: nutrition

INTERVENTIONS:
Other: nutrition — type and amount of food eaten or type of oral nutritional supplements as well as enteral or parenteral nutrition
  Other Names: hospital food; oral protein energy supplements; enteral nutrition; parenteral nutrition

SUMMARY:
Malnutrition at hospital admission is a risk factor for an unfavourable outcome, prolonged hospital stay and delayed recovery. In these patients the incidence of complications such as nosocomial infections, poor ventilatory function, prolonged bed rest is increased. In addition a relevant proportion of patients have a nutritional intake below their needs during hospitalisation.Mortality has been shown to be up to 8 times higher and dependency at discharge up to 3 times more frequent when actual food intake was below 25% of calculated needs.

The aim of this international cross-sectional multicentre audit and registry is to generate a risk and level of nutritional intervention profile for an individual unit/ward based on case-mix, nutrition care and available structures. This profile should give a snapshot on the relation of risk to resource allocation. The audit is unit centered. Each unit gets as a feedback anonymously its position compared with all other participating units. Risk adjustment for selected patient groups, social environments and structures is planned.

In conclusion this audit/registry will serve five distinct aims:

* Generate a precise map of the prevalence of malnutrition before admission and of decreased nutrient intake according to risk factors, medical specialty, organisational structures and countries.
* Increase in awareness for clinical nutrition in patients, caregiver and hospital managers.
* Enlarge and maintain a reference database for hospitalised patients
* Provide individual unit benchmarking

DETAILED DESCRIPTION:
One day international cross-sectional audit in all types of hospital wards. Intensive care units are excluded. Data are collected with the help of questionnaires. Anonymised data entry into the audit database is done with individual and anonymous center and unit-codes.

The data collected consist of four parts:

1. Unit organisation and structures:

   Structural information about the unit (one sheet / unit) to be filled by the unit supervising physician together with the nursing head.
2. Patient's demographics & medical information:

   Demographic profile, diagnostic category based on ICD 10 and nutritional interventions for all patients (one line / patient) to be filled by a responsible person from the medical staff. Oncological patients have an additional caregiver sheet to define precisely cancer stage and specific treatment.
3. Individual self-administered patient questionnaire:

   Each patient should document her/his nutritional intake during the study period. In addition patients may be asked to fill a questionnaire about changes in nutritional habits and reasons for decreased nutritional intake from the patient's perspective. Oncological patients have an additional optional patient sheet to determine the specific nutritional problems and supportive treatments used.
4. Individual patient outcome:

hospital cohort: at hospital discharge or day 30, whatever comes first: date of unit discharge, date of hospital discharge, site of discharge and health status.

Participation rules:

1. A user needs to register to nutritionDay as a member to the nutritionDay network. Each may choose a personal user name. Each user needs to provide a valid email address. After responding to a validation email the user is registered with the chosen user name. User details are stored on a system that is not connected to the nutritionDay registry at any time. One user may serve as contact for several units and centers.
2. A user may order codes for participation for one or several centers and units. Access to the registry is only possible with a center code and unit code. These codes are selected from a list of random numbers.

Audit/registry recruitment plan:

Participation to the registry is voluntary. There is actually no participation fee. All necessary information can be obtained from a dedicated website (www.nutritionday.org). Participation can be promoted via international and national scientific societies, universities, health care organisations or governmental agencies as well as via advertisement at international and national congresses. The target would be all types of hospital wards within hospitals of different sizes and level of care.

Risk and benefit assessment:

The benefit for each patient is that awareness and knowledge about nutrition related factors and treatment options in the treating unit is increased. There is no individual risk since the audit is purely observational.

The benefit for the individual unit is to receive an extensive benchmarking report displaying the unit data in comparison with all units from the same specialty from the previous 3 years immediately after the end of data entry and a validation step. Units or groups of units may request specific reports that can be obtained only after a case by case agreement and financial coverage. All data used as a reference for benchmarking purpose are from units where a minimum of 60% of actually present patients have been recruited and the outcome at day 30 is available in more than 80% of these patients. There is no risk for the unit since anonymity of unit is structurally strictly maintained.

The benefit for the registry up-to-date data enabling benchmarking in pace with medical and care evolution. Moreover the registry data are used for research of the scientific community.

The aim is to recruit a minimum of 10-50 units with 20-30 beds per participating country. A minimum of 10 units per medical specialty will be necessary to allow specialty adjustment.

Data security:

On the datasheets the unit and the hospital/center are identified by a numeric code delivered after application to the nutritionDay coordinating center by an automatic system. The only requirement is a valid email address for direct communication with the unit.

Patients are usually identified on the locally used questionnaires by initials and age, but use of initials is not mandatory. Consecutive numbering is also possible. Only the participating unit has to trace patients identifier to be able to collect hospital outcome at day 30 after nutritionDay and to answer automatic requests for data clarification during the data quality feedback.

During data entry into the electronic registry only anonymous codes for center, unit and patients are possible. Thus the data handling centre cannot trace data back to an individual patient. The access to data entry is protected by anonymous center-code and unit-code.

Typically all data are collected via a dedicated website accessed via www.nutritionday.org .

The protected data server is run by the Center for Medical Statistics Informatics and Intelligent Systems (CEMSIS) of the Medical University Vienna. The data server is mirrored and backed up. The data server is protected within the University Firewall against external access.

Data feedback and individual unit report

All participating units are entitled to receive a bench-marking report from the registry. The report generator is started by the participating unit, when data entry has been completed. As a first step each unit receives a data feedback sheet that is based on an electronic data plausibility and missing data analysis. After stating that all data are correctly entered the final report can be generated. This final report offers complete descriptive statistics of the unit data compared to the reference data from the previous 4 years of the corresponding specialty. Only data from units fulfilling a high data quality standard are used for the reference. More than 60% of the patients present in the unit need to participate and 80% of these patients need to have their outcome recorded. Optionally the period used for comparison can be extended until 2006. All descriptive statistics represent prevalent data and are not corrected for cross-sectional sampling to allow direct data control and interpretation.

All downloaded reports of a unit are consecutively numbered and stored for documentation purpose.

Data analysis and modelling:

The first aim of the project is to serve local specialty specific and up-to-date benchmarking with regard nutrition and feeding status , risk profile and nutrition care. Given the typical cross-sectional sample of 20-30 patients frequent risk factors can be easily compared because such risk factors as recent weight loss or less than normal eating are observed in one third to half of the patients.

The second aim is scientific data analysis. The actual research questions are:

* Identifying the risk factors associated with decreased eating.
* Analysing the impact of risk factors for increased length of hospital stay
* Analysing time-trends in risk profile and nutrition care
* Analysing the economic impact of nutrition risk factors on the health care system
* Updating the PANDORA score if major change in performance is identified

The actual database includes 103 920 patients for the period 2006-2012 and allow the following precision for estimating the prevalence of risk factors:

Risk factor prevalence 1% precision as 95% CI 0.93-1.07%

Risk factor prevalence 5% precision as 95% CI 4.87-5.14%

Risk factor prevalence 10% precision as 95% CI 9.81-10.19%

Risk factor prevalence 20% precision as 95% CI 19.75-20.25%

Risk factor prevalence 30% precision as 95% CI 29.72-30.29%

Risk factor prevalence 40% precision as 95% CI 39.70-40.30%

Given the typical participation of 12 000-20 000 patients annually, the investigators expect to have a sufficiently precise database for benchmarking, when using the last 4 years data.

For the scientific data analysis the investigators use COX-regression or general linear model with proper weighting of observations to account for the effect of cross-sectional sampling for events such as discharge or death and linear regression models to analyse length of stay. Whenever several events can occur in a patient a competing risk analysis is performed.

All data analysis will be done at the Dept. for Medical Statistics, Medical University Vienna. After publication of the multinational results, all national datasets will be available for national publication based on a research plan, if the number of wards is large enough to ensure anonymity for the individual ward within the country.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in a given ward and present within the unit from 7H00 to 19H00 (e.g.) during the first nursing shift of the nutritionDay (one given day per year), including admissions and discharges within the period.

Questionnaire especially dedicated to children and young adults are provided for patients aged 7-17. Questionnaires for children can be completed by the patients themselves or by a legal guardian.

* Patients may accept to participate only for the medical documentation part from the caregiver sheet (sheet 2) and individual patient outcome (sheet 4), but refuse to fill the individual patient questionnaire (sheet 3).

Exclusion Criteria:

* Patient with an age < 6 a.
* Patients unable to understand and answer questions because none of the 31 available languages is understood for the hospital cohort.
* Patient's refusal to answer the patient specific questionnaire or refusal of medical data use for auditing and research.
* Patients admitted and discharged during the same calendar day.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients hospitalised on a given day in hospital wards.
Sampling Method: Non-Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2006-01; Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
mortality in hospital (hospital cohort) | 30 days
  date of death within 30 days of sampling day

SECONDARY OUTCOMES:
length of hospital stay | 30 days
  date of discharge or death within 30 days after the cross-sectional sampling day

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Hiesmayr, MD, MSc, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna, CEMSIIS, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Upon submission of a research proposal data anonymised data are shared with researcher. Each proposal is submitted to the supervisory board for approval.
Supporting Information: Study Protocol, ICF
Time Frame: 1 month
Access Criteria: submission of a research proposal and approval by the scientific committee of nutritionDay as well as a data sharing contract according to Medical University Legal Department

REFERENCES:
- [Background] Frantal S, Pernicka E, Hiesmayr M, Schindler K, Bauer P. Length bias correction in one-day cross-sectional assessments - The nutritionDay study. Clin Nutr. 2016 Apr;35(2):522-527. doi: 10.1016/j.clnu.2015.03.019. Epub 2015 Apr 7. PMID 25912233
- [Result] Hiesmayr M, Schindler K, Pernicka E, Schuh C, Schoeniger-Hekele A, Bauer P, Laviano A, Lovell AD, Mouhieddine M, Schuetz T, Schneider SM, Singer P, Pichard C, Howard P, Jonkers C, Grecu I, Ljungqvist O; NutritionDay Audit Team. Decreased food intake is a risk factor for mortality in hospitalised patients: the NutritionDay survey 2006. Clin Nutr. 2009 Oct;28(5):484-91. doi: 10.1016/j.clnu.2009.05.013. Epub 2009 Jul 1. PMID 19573957
- [Result] Schindler K, Pernicka E, Laviano A, Howard P, Schutz T, Bauer P, Grecu I, Jonkers C, Kondrup J, Ljungqvist O, Mouhieddine M, Pichard C, Singer P, Schneider S, Schuh C, Hiesmayr M; NutritionDay Audit Team. How nutritional risk is assessed and managed in European hospitals: a survey of 21,007 patients findings from the 2007-2008 cross-sectional nutritionDay survey. Clin Nutr. 2010 Oct;29(5):552-9. doi: 10.1016/j.clnu.2010.04.001. PMID 20434820
- [Result] Lainscak M, Farkas J, Frantal S, Singer P, Bauer P, Hiesmayr M, Schindler K. Self-rated health, nutritional intake and mortality in adult hospitalized patients. Eur J Clin Invest. 2014 Sep;44(9):813-24. doi: 10.1111/eci.12300. PMID 25039263
- [Result] Hiesmayr M, Frantal S, Schindler K, Themessl-Huber M, Mouhieddine M, Schuh C, Pernicka E, Schneider S, Singer P, Ljunqvist O, Pichard C, Laviano A, Kosak S, Bauer P. The Patient- And Nutrition-Derived Outcome Risk Assessment Score (PANDORA): Development of a Simple Predictive Risk Score for 30-Day In-Hospital Mortality Based on Demographics, Clinical Observation, and Nutrition. PLoS One. 2015 May 22;10(5):e0127316. doi: 10.1371/journal.pone.0127316. eCollection 2015. PMID 26000634
- [Result] Cereda E, Klersy C, Hiesmayr M, Schindler K, Singer P, Laviano A, Caccialanza R; NutritionDay Survey Collaborators. Body mass index, age and in-hospital mortality: The NutritionDay multinational survey. Clin Nutr. 2017 Jun;36(3):839-847. doi: 10.1016/j.clnu.2016.05.001. Epub 2016 May 15. PMID 27236599
- [Derived] Moick S, Hiesmayr M, Mouhieddine M, Kiss N, Bauer P, Sulz I, Singer P, Simon J. Reducing the knowledge to action gap in hospital nutrition care - Developing and implementing nutritionDay 2.0. Clin Nutr. 2021 Mar;40(3):936-945. doi: 10.1016/j.clnu.2020.06.021. Epub 2020 Jul 2. PMID 32747205
- [Derived] Moick S, Simon J, Hiesmayr M. Nutrition care quality indicators in hospitals and nursing homes: A systematic literature review and critical appraisal of current evidence. Clin Nutr. 2020 Jun;39(6):1667-1680. doi: 10.1016/j.clnu.2019.07.025. Epub 2019 Aug 7. PMID 31447247
- [Derived] Schindler K, Themessl-Huber M, Hiesmayr M, Kosak S, Lainscak M, Laviano A, Ljungqvist O, Mouhieddine M, Schneider S, de van der Schueren M, Schutz T, Schuh C, Singer P, Bauer P, Pichard C. To eat or not to eat? Indicators for reduced food intake in 91,245 patients hospitalized on nutritionDays 2006-2014 in 56 countries worldwide: a descriptive analysis. Am J Clin Nutr. 2016 Nov;104(5):1393-1402. doi: 10.3945/ajcn.116.137125. Epub 2016 Oct 12. PMID 27733401
- See also: official registry website — http://www.nutritionday.org